CLINICAL TRIAL: NCT02520921
Title: Aspirin With a Novel Twice-a-day Administration in Diabetic Patients With Acute Coronary Syndrome to Minimize Recurrence of Acute Ischemic Events or New Urgent Revascularization
Brief Title: Aspirin Twice a Day in Patients With Diabetes and Acute Coronary Syndrome
Acronym: ANDAMAN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P141005; 2015-000947-18 (EudraCT Number)
Record Dates: First submitted 2015-06-12; First posted 2015-08-13 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Diabetes Mellitus; Acute Coronary Syndrome; Coronary Artery Disease; Obesity
Keywords: Diabetes mellitus; Acute coronary syndrome; Coronary artery disease; Aspirin; Secondary prevention; Obesity
MeSH Terms: conditions — Diabetes Mellitus; Acute Coronary Syndrome; Coronary Artery Disease; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 : Novel strategy (Active Comparator): enteric coated aspirin 100 mg in the morning and 100 mg in the evening
  Interventions: Drug: Novel strategy Aspirin
- Arm 2 : Conventional strategy (Active Comparator): enteric coated aspirin 100 mg in the morning
  Interventions: Drug: Conventional strategy Aspirin

INTERVENTIONS:
Drug: Novel strategy Aspirin — Aspirin twice a day : enteric coated enteric coated aspirin given twice a day, 100 mg in the morning and 100 mg in the evening (i.e. 200mg/day)
  Arms: Arm 1 : Novel strategy
Drug: Conventional strategy Aspirin — Aspirin once day: enteric coated aspirin 100 mg in the morning (i.e. 100mg/day)
  Arms: Arm 2 : Conventional strategy

SUMMARY:
To compare treatment with Aspirin Protect® twice a day (100 mg in the morning and 100 mg in the evening) versus Aspirin Protect® 100 mg once per day on a composite end-point of ischemic events in diabetic patients, or in patients with a known risk factor for non-optimal aspirin response (obesity, abdominal obesity or coronary event occurring with long-term aspirin),with acute coronary syndrome. It is expected that aspirin taken twice a day will reduce the occurrence of new ischemic event after acute coronary syndrome in diabetic patients or in patients with a known risk factor.

DETAILED DESCRIPTION:
Patients who show high persistent platelet reactivity under aspirin are increasingly becoming an issue of clinical concern. Several studies have suggested that giving aspirin more frequently is very effective for reducing aspirin high persistent platelet reactivity, especially in diabetic patientsor in patients with a known risk factor. The aim of the study is to evaluate low dose of aspirin twice a day (compared to once a day) for the reduction of ischemic events in diabetic patients or in patients with a known risk factor, with acute coronary syndrome.

Experimental Design:

A multicenter, randomised, parallel group comparing aspirin given twice a day compared to once per day in diabetic patients, or in patients with a known risk factor for non-optimal aspirin response (obesity, abdominal obesity or coronary event occurring with long-term aspirin),with acute coronary syndrome.

Primary objective:

To compare treatment with Aspirin Protect® twice a day (100 mg in the morning and 100 mg in the evening) versus Aspirin Protect® 100 mg once per day on a composite end-point of ischemic events in diabetic patients, or in patients with a known risk factor for non-optimal aspirin response (obesity, abdominal obesity or coronary event occurring with long-term aspirin),with acute coronary syndrome.

Secondary objectives:

* To compare treatment with Aspirin Protect® twice a day (100 mg in the morning and 100 mg in the evening) versus Aspirin Protect® 100 mg once per day on net clinical benefit combining the ischemic and bleeding events in diabetic patients, or in patients with a known risk factor for non-optimal aspirin response (obesity, abdominal obesity or coronary event occurring with long-term aspirin),with acute coronary syndrome.
* To compare treatment with Aspirin Protect® twice a day (100 mg in the morning and 100 mg in the evening) versus Aspirin Protect® 100 mg once per day on cardiac events in diabetic patients, or in patients with a known risk factor for non-optimal aspirin response (obesity, abdominal obesity or coronary event occurring with long-term aspirin),with acute coronary syndrome.
* To compare treatment with Aspirin Protect® twice a day (100 mg in the morning and 100 mg in the evening) versus Aspirin Protect® 100 mg once per day in each of individual component of the main criterion.
* To confirm the safety of the innovative strategy (aspirin twice a day) concerning major bleeding events.

Study enrollment:

Multicentric national study involving 42 centers in France The duration is expected to be 24 months of recruitment. Patients will be randomized during the index hospitalization for acute coronary syndrome and before discharge between a conventional strategy of enteric coated aspirin 100mg per day with the standard of care or a innovative strategy of enteric coated aspirin 100mg morning and evening. Patients will be followed at one month, six months, one year and 18 months

Statistical analysis:

The study will include 2574 patients. We hypothesized that at 18 months, there will be an event rate of 22% for "death, MI, stroke, urgent revascularization, or acute arterial thrombotic event in the group treated with aspirin and we expect a decrease of the primary event of 20% (relative variation) using aspirin twice a day corresponding to an event rate of 17.6%.

A sample size of 1287 patients /group will allow an 80% power to detect this difference using a log-rank test at a two-sided 5% significance level. The study will include 2574 diabetic patients, or patients with a known risk factor for non-optimal aspirin response.

The primary analysis is based on the Intention To Treat population and the primary endpoint. The primary analysis on the primary endpoint will be carried out using a log-rank test for survival analysis. The 95% confidence interval of the hazard ratio will be presented. In addition the survival status during 18 months follow-up will be described by showing Kaplan-Meier curves.

Primary outcome according to pre-specified subgroups:

* Age: patients < 75 years or patient ≥75 years
* Gender: male or female
* Insulin vs no insulin treatment
* Type of acute coronary syndrome : STEMI vs NSTEMI
* Type of ADP inhibitor cotreatment
* Treatment strategy medical vs invasive (angioplasty or CABG surgery)
* Peripheral artery disease Yes/No
* GRACE score > or ≤140
* Left ventricular ejection fraction > or ≤ 40%
* Prior stroke Yes/No
* previous treatment with aspirin Yes/No
* initial HbA1C level > or ≤8%
* duration of diabetes > or ≤10 years
* Weight <60; 60-90; >90kg
* PPI use Yes/No

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus defined as (≥ 1 item)

  * Treated diabetes mellitus
  * 2 fasting glucose levels ≥ 7 mmol/l after admission
  * glucose level ≥ 11 mmol/l after admission (any moment)
  * HbA1C ≥ 6.5% OR
* Factor of aspirin lack of efficacy defined as (≥ 1 item)

  * Obesity defined as BMI≥27kg/m2
  * Waist circumference ≥ 88cm for women or ≥102cm for men
  * Index event occurring under chronic low dose of aspirin (<300mg)

AND

- Acute coronary syndrome defined as:

* Acute coronary syndrome with ST-segment elevation (STEMI) is defined as chest pain (≥ 30min) with persistent ST-segment elevation in at least two contiguous leads (≥1mm) or a new left bundle-branch block and the intention to perform primary PCI or thrombolysis.
* Acute coronary syndrome without ST-segment elevation (NSTEMI) is defined as universal myocardial definition:

Detection of cardiac biomarker values elevation [preferably cardiac troponin (cTn)] with at least one value above the 99th percentile upper reference limit (URL) and with at least one of the following:

* Symptoms of ischemia
* New or presumed new significant ST-segment-T wave (ST-T) changes except ST elevation
* Development of pathological Q waves in the ECG
* Imaging evidence of new loss of viable myocardium or new regional wall motion abnormality
* Identification of an intracoronary thrombus by angiography

  * included after the angiography showing stenosis ≥50% and before discharge
  * signed informed consent and ≥18 years old

Exclusion Criteria:

* Allergy or contraindication to aspirin (Hypersensitivity to aspirin or any of the excipients, history of asthma induced by the administration of salicylates, ongoing peptic ulcer, constitutional or acquired haemorrhagic disease including gastrointestinal bleeding, history of hemorrhagic stroke and thrombocytopenia, pregnancy after 24 weeks of gestation, risk of bleeding, severe renal failure, severe hepatic impairment, uncontrolled severe heart failure
* Concomitant anticoagulation therapy that cannot be stopped
* Fibrinolytic therapy less than 24 hours.
* Unstable patients according to investigator: use of amine or mechanical device (IABP, ECMO or similar) or mechanical ventilation during index hospitalization
* Index event is an acute complication of coronary revascularization (PCI or CABG)
* Known serious hematological disorder
* Proven gastric or duodenal ulcer in the past 3 months
* Previous hemorrhagic stroke, previous cranial bleeding, intracranial neoplasia, arterio-venous malformation
* Any condition that may put the patient at risk or influence study result in the investigators' opinion (active cancer ….) or that increase the risk for non-compliance or being lost to follow-up
* Concomitant treatment with methotrexate or with chronic non-steroidal anti-inflammatory drug
* Pregnancy or lactation or woman of childbearing age without contraception
* Participant in an another investigational drug study within 30 days
* Patients under curatorship
* No social security

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2484 (Actual)
Dates: Start 2016-06-13 (Actual); Primary Completion 2024-07-18 (Actual); Study Completion 2024-07-18 (Actual)

PRIMARY OUTCOMES:
first main vascular event occurring within the 18 months after randomization among the following: Death (any), Myocardial infarction, Stroke, Urgent coronary revascularization and/or stent thrombosis, Acute arterial thrombotic event | at18 months

SECONDARY OUTCOMES:
Major bleeding (type 3 to 5 following BARC classification | at18 months
Net clinical benefit: Death (any), Myocardial infarction, Stroke, Urgent coronary revascularization and/or stent thrombosis, Acute arterial thrombotic event, Major bleeding | at18 months
Cardiac endpoint: Cardiovascular death / Myocardial infarction | at18 months
Death, myocardial infarction, stroke, urgent revascularization, stent thrombosis, acute arterial thrombotic event and major bleeding analyzed specifically and separately | at18 months

CONTACTS AND LOCATIONS:
Overall Officials: Patrick HENRY, MD, PhD, Principal Investigator — Assistance Publique
Locations (1):
- Department of Cardiology - Lariboisiere Hospital, Paris, France

REFERENCES:
- [Derived] Dillinger JG, Pezel T, Batias L, Angoulvant D, Goralski M, Ferrari E, Cayla G, Silvain J, Gilard M, Lemesle G, Souteyrand G, Lim P, Roubille F, Georges JL, Bal Dit Sollier C, Petroni T, Morel O, Delarche N, Elbaz M, Puymirat E, Toupin S, Montalescot G, Drouet L, Vicaut E, Henry P; ANDAMAN Investigators of the ACTION Study Group. Aspirin dosing after acute coronary syndrome with suspected aspirin resistance: the ANDAMAN trial. Eur Heart J. 2025 Aug 30:ehaf680. doi: 10.1093/eurheartj/ehaf680. Online ahead of print. PMID 40884757
- [Derived] Dillinger JG, Pezel T, Batias L, Angoulvant D, Goralski M, Ferrari E, Cayla G, Silvain J, Gilard M, Lemesle G, Souteyrand G, Lim P, Roubille F, Georges JL, Bal Dit Sollier C, Petroni T, Morel O, Delarche N, Elbaz M, Puymirat E, Toupin S, Montalescot G, Drouet L, Vicaut E, Henry P; ANDAMAN Investigators of the ACTION Study Group. Twice-a-day administration of aspirin in patients with diabetes mellitus or aspirin resistance after acute coronary syndrome: Rationale and design of the randomized ANDAMAN trial. Am Heart J. 2025 Oct;288:101-110. doi: 10.1016/j.ahj.2025.04.016. Epub 2025 Apr 21. PMID 40268181